CLINICAL TRIAL: NCT05115578
Title: Remifentanil Pharmacodynamics During Conscious Sedation From the Algometry Perspective. An Essential Standpoint to be Considered in Opioids Time-course Modelling Validation
Brief Title: Remifentanil Effect-site Prediction by Algometry
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: EPA (AG) 33/2017 (5097)
Record Dates: First submitted 2021-09-15; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Conscious Sedation Failure During Procedure
Keywords: Remifentanil; Algometry; Pharmacodynamics; TCI Infusion system; Conscious Sedation
MeSH Terms: interventions — Remifentanil; Injections; Analgesics, Opioid; Midazolam; Benzodiazepines; Saline Solution; Sodium Chloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I TCI effect-site target infusion of 1.5 ng/ml of remifentanil: Group I of 35 patients received a constant TCI effect-site target infusion of 1.5 ng/ml of remifentanil for 25 min.
  Interventions: Drug: Remifentanil 1 MG Injection [Ultiva]; Device: Algometry
- Group II TCI effect-site target infusion of 1.5 ng/ml of remifentanil + 1 mg Midazolam iv: Group II of 35 patients received a constant TCI effect-site target infusion of 1.5 ng/ml of remifentanil for 25 min with a bolus of 1 mg of midazolam previous to the remifentanil infusion
  Interventions: Drug: Remifentanil 1 MG Injection [Ultiva]; Drug: Midazolam 1 MG/ML Prefilled Syringe; Device: Algometry
- Group III Control: Group III of 30 patients. The same TCI system provided the saline solution in the control group under an equivalent simulation profile to the remifentanil administration
  Interventions: Drug: Saline solution; Device: Algometry

INTERVENTIONS:
Drug: Remifentanil 1 MG Injection [Ultiva] — Group I TCI effect-site target infusion of 1.5 ng/ml of remifentanil.
  Other Names: Opioid
  Groups: Group I TCI effect-site target infusion of 1.5 ng/ml of remifentanil; Group II TCI effect-site target infusion of 1.5 ng/ml of remifentanil + 1 mg Midazolam iv
Drug: Midazolam 1 MG/ML Prefilled Syringe — Group II TCI effect-site target infusion of 1.5 ng/ml of remifentanil + 1 mg Midazolam iv
  Other Names: Benzodiazepine
  Groups: Group II TCI effect-site target infusion of 1.5 ng/ml of remifentanil + 1 mg Midazolam iv
Drug: Saline solution — Group III Control
  Other Names: 0.9% Sodium Chloride Injection
  Groups: Group III Control
Device: Algometry — The algometry technique is used to assess the pain pressure threshold as an analgesic effect of remifentanil concerning Minto's model prediction.
  Other Names: Somedic Type II®, Sweden

SUMMARY:
This study validates the pharmacodynamic analgesic predictions (effect) given by Minto's remifentanil pharmacokinetic and dynamic model in conscious sedation. This standard model is based on the electroencephalogram (EEG) changes induced by this opioid as a proxy for describing the remifentanil analgesic effect, which might be only valid for high concentrations. Validation of the standard remifentanil model for low concentrations under sedation is needed for safer remifentanil administration.

DETAILED DESCRIPTION:
According to pharmacokinetic and-dynamic (PK/PD) models, the proper use of anesthetics depends on the effect-sites mechanisms and the time-courses of action. This aspect is crucial for the practitioners to target the desired effect-site concentrations of the drugs (drug concentration at brain) by optimizing the drug administration using target control infusion (TCI) systems operating under these model predictions.

For more than two decades, the pharmacodynamic properties of remifentanil relied on Minto's model, which is based on processed EEG as the reference to quantify the analgesic effect and effect-site concentration estimate. This remifentanil pharmacodynamic was modeled under conditions administered to volunteers rapidly and at very high doses to induce substantial changes in the spontaneous processed EEG. The experimental concentrations and infusion rates are far from sedative levels, where the EEG has shown a clear response to hypnosis but not to analgesia or nociception.

Under the hypothesis that pharmacological models should predict equally well the effects induced by drugs at different concentrations levels, the purpose of this study is to evaluate and validate the pharmacodynamic predictions given by Minto's model in patients under conscious sedation using the algometry as a reference of nociception.

The study recruits 100 female patients scheduled for benign gynecological surgery divided into three groups. A group of 35 patients receives a constant TCI effect-site target infusion of 1.5 ng/ml of remifentanil for 25 min. The second group of 35 follow the same protocol with a bolus of 1 mg of midazolam before the remifentanil infusion. The rest configures the control group under saline solution.

Experimental data consist of basal algometry (pressure pain threshold) aside from BIS index, blood pressure, and heart rate values and at time-points of 1.5, 5, 10, 15, 18, 20, and 25 minutes after induction.

Minto's remifentanil pharmacodynamic model validation relies on comparing the levels and temporal evolution of the algometry measurements during the whole experiment concerning the effect-site estimations provided by the TCI-pump Minto's model.

ELIGIBILITY:
Inclusion Criteria:

* Female patients scheduled for benign gynaecological surgery
* 18-80 years old
* ASA I-III

Exclusion Criteria:

* Morbid obesity
* Conduct disorder or anxiety-depressive syndrome
* Chronic treatment with psychotropic drugs or opiates
* Pregnancy
* Alcohol abuse
* Documented allergy to remifentanil or midazolam
* Refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We enrolled 100 female patients scheduled for benign gynaecological surgery. A group of 35 patients received a constant TCI effect-site target infusion of 1.5 ng/ml of remifentanil for 25 min. The second group of 35 followed the same protocol with a bolus of 1 mg of midazolam previous to the remifentanil infusion to evaluate potential anxiolysis effects. The rest configured to the control group.
  Algometry was used to quantify pressure pain thresholds regarding basal measurements at time-points of 1.5, 5, 10, 15, 18, 20, and 25 min after induction began beside the blood pressure and heart rate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold (PPT) Baseline | Baseline
  Measurement of pressure pain threshold (0 - 1.000 kPa) by algometry before starting the administration of remifentanil.
Pressure pain threshold (PPT) 1.5 minutes | 1.5 minutes
  Measurement of pressure pain threshold (0 - 1.000 kPa) by algometry 1.5 minutes after starting the administration of remifentanil.
Pressure pain threshold (PPT) 5 minutes | 5 minutes
  Measurement of pressure pain threshold (0 - 1.000 kPa) by algometry 5 minutes after starting the administration of remifentanil.
Pressure pain threshold (PPT) 10 minutes | 10 minutes
  Measurement of pressure pain threshold (0 - 1.000 kPa) by algometry 10 minutes after starting the administration of remifentanil.
Pressure pain threshold (PPT) 15 minutes | 15 minutes
  Measurement of pressure pain threshold(0 - 1.000 kPa) by algometry 15 minutes after starting the administration of remifentanil.
Pressure pain threshold (PPT) 18 minutes | 18 minutes
  Measurement of pressure pain threshold (0 - 1.000 kPa) by algometry 18 minutes after starting the administration of remifentanil.
Pressure pain threshold (PPT) 20 minutes | 20 minutes
  Measurement of pressure pain threshold (0 - 1.000 kPa) by algometry 20 minutes after starting the administration of remifentanil.
Pressure pain threshold (PPT) 25 minutes | 25 minutes
  Measurement of pressure pain threshold (0 - 1.000 kPa) by algometry 25 minutes after starting the administration of remifentanil.
Infusion rate | Continous measurements every 1 second for the whole experiment of 25 minutes
  Remifentanil infusion rate (ml/h) administered during the experiment to the patient provided by the TCI system.
Remifentanil Plasma Concentration (Cp) | Continous measurements every 1 second for the whole experiment of 25 minutes
  Patient's remifentanil plasma concentration (ng/ml) evolution during the experiment given by Minto's model implemented in the TCI system.
Remifentanil Effect Concentration (Ce) | Continous measurements every 1 second for the whole experiment of 25 minutes
  Patient's remifentanil effect concentration (ng/ml) evolution during the experiment given by Minto's model implemented in the TCI system.

SECONDARY OUTCOMES:
Age | Single annotation.
  Apart from standard anthropometric data (Weight, Height, etc), age is of significant relevance for evaluating the possible effect of age on the pharmacodynamic properties of remifentanil and the algometry.
Mean arterial pressure (MAP) Baseline | Baseline
  Baseline mean arterial pressure (mmHg) from standard hemodynamic monitor.
Mean arterial pressure (MAP) 1.5 min | 1.5 minutes
  Measurement of mean arterial pressure (mmHg) 1.5 minutes after starting the administration of remifentanil.
Mean arterial pressure (MAP) 5 min | 5 minutes
  Measurement of mean arterial pressure (mmHg) 5 minutes after starting the administration of remifentanil.
Mean arterial pressure (MAP) 10 min | 10 minutes
  Measurement of mean arterial pressure (mmHg) 10 minutes after starting the administration of remifentanil.
Mean arterial pressure (MAP) 15 min | 15 minutes
  Measurement of mean arterial pressure (mmHg) 15 minutes after starting the administration of remifentanil.
Mean arterial pressure (MAP) 18 min | 18 minutes
  Measurement of mean arterial pressure (mmHg) 18 minutes after starting the administration of remifentanil.
Mean arterial pressure (MAP) 20 min | 20 minutes
  Measurement of mean arterial pressure (mmHg) 20 minutes after starting the administration of remifentanil.
Mean arterial pressure (MAP) 25 min | 25 minutes
  Measurement of mean arterial pressure (mmHg) 25 minutes after starting the administration of remifentanil.
Heart Rate (HR) Baseline | Baseline
  Baseline measurement of heart rate (beats/min)
Heart Rate (HR) 1.5 min | 1.5 minutes
  Measurement of heart rate (beats/min) 1.5 minutes after starting the administration of remifentanil.
Heart Rate (HR) 5 min | 5 minutes
  Measurement of heart rate (beats/min) 5 minutes after starting the administration of remifentanil.
Heart Rate (HR) 10 min | 10 minutes
  Measurement of heart rate (beats/min) 10 minutes after starting the administration of remifentanil.
Heart Rate (HR) 15 min | 15 minutes
  Measurement of heart rate (beats/min) 15 minutes after starting the administration of remifentanil.
Heart Rate (HR) 18 min | 18 minutes
  Measurement of heart rate (beats/min) 18 minutes after starting the administration of remifentanil.
Heart Rate (HR) 20 min | 20 minutes
  Measurement of heart rate (beats/min) 20 minutes after starting the administration of remifentanil.
Bispectrum (BIS) Baseline | Baseline
  Baseline measurement of EEG Bispectral index (adimensional index from 0- to 100).
Bispectrum (BIS) 1.5 minutes | 1.5 minutes
  EEG Bispectral index (adimensional index from 0- to 100) 1.5 minutes after starting the administration of remifentanil.
Bispectrum (BIS) 5 minutes | 5 minutes
  EEG Bispectral index (adimensional index from 0- to 100) 5 minutes after starting the administration of remifentanil.
Bispectrum (BIS) 10 minutes | 10 minutes
  EEG Bispectral index (adimensional index from 0- to 100) 10 minutes after starting the administration of remifentanil.
Bispectrum (BIS) 15 minutes | 15 minutes
  EEG Bispectral index (adimensional index from 0- to 100) 15 minutes after starting the administration of remifentanil.
Bispectrum (BIS) 20 minutes | 20 minutes
  EEG Bispectral index (adimensional index from 0- to 100) 20 minutes after starting the administration of remifentanil.
Bispectrum (BIS) 25 minutes | 25 minutes
  EEG Bispectral index (adimensional index from 0- to 100) 25 minutes after starting the administration of remifentanil.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Abad-Torrent, M.D, Principal Investigator — University Vall d'Hebron Hospital
Locations (1):
- Ana Abad-Torrent, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided